CLINICAL TRIAL: NCT01367613
Title: A Three-Month Open-Label Treatment Extension of Protocol MNTX 302
Brief Title: Open-Label Treatment Extension of Protocol MNTX 302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 302EXT
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Terminal Illness
Keywords: Advanced medical illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone

INTERVENTIONS:
Drug: SC Methylnaltrexone

SUMMARY:
This is a 3 month open-label extension study that allows patients who completed Protocol MNTX 302 to receive SC MNTX.

ELIGIBILITY:
Inclusion Criteria:

1. Must be enrolled and consented within 28 days of the end of study visit of MNTX 302 and 14 or more days from first dose of study drug in MNTX 302.
2. Negative pregnancy test
3. Stable vital signs

Exclusion Criteria:

1. Women who are pregnant and/or nursing
2. Received any investigational product, other than MNTX, in the past 30 days
3. Evidence of fecal impaction
4. Clinically significant active diverticular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 3 months
  To provide access to treatment with MNTX, administered SC, to patients who completed Progenics' Protocol MNTX 302

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States